CLINICAL TRIAL: NCT03746392
Title: Using the Electronic Health Record to Identify and Promote Goals-of-Care Communication
Brief Title: Project to Improve Communication About Serious Illness - Pilot Study
Acronym: PICSI-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, R. Engelberg, ResearchProfessor, Department of Medicine, SOM: Department of Medicine: Pulmonary, Critical Care and Sleep Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00004821
Record Dates: First submitted 2018-11-09; First posted 2018-11-19 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Malignant Neoplasm; Leukemia, Lymphocytic, Chronic, B-Cell; Lung Disease Chronic; Congestive Heart Failure; Liver Failures, Chronic; Renal Insufficiency, Chronic; Dementia; Diabetes Complications; Peripheral Vascular Disease; Frail Elderly
MeSH Terms: conditions — Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Heart Failure; End Stage Liver Disease; Renal Insufficiency, Chronic; Dementia; Diabetes Complications; Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jumpstart Intervention (Experimental)
  Interventions: Behavioral: Jumpstart Intervention
- Usual Inpatient Hospital Care (No Intervention)

INTERVENTIONS:
Behavioral: Jumpstart Intervention — The intervention has 4 steps: use electronic medical record (EHR) to identify seriously ill, hospitalized patients with no documentation of a goals-of-care (GOC) discussion during their current admission; the enrolled patient or his/her surrogate completes a survey assessing preferences for discussions about GOC, barriers to having such discussions, and current GOC which is used to create a "Jumpstart" form designed to prompt and guide a GOC discussion between the patient or surrogate and the clinicians caring for the patient; use natural language processing/machine learning (NLP/ML) approach to identify GOC discussions or advance directives in the EHR that occurred prior to admission and include this information on the Jumpstart form; and, deliver the Jumpstart form to the primary clinician team. The patient or surrogate is also provided with a version of the form.
  Arms: Jumpstart Intervention

SUMMARY:
This two-year pilot study will test whether a one-page "Jumpstart Form" will affect goals-of-care discussions in the hospital. This form will be provided to clinicians and will include patient-specific information about preferences for goals-of-care communication and for care, as well as tips to improve this communication. Jumpstart forms will also be provided to patients or, if they are unable to communicate, their surrogates/family members. The information on the form will be obtained from questionnaires. The form is tailored to help patients and surrogates talk with clinicians about goals of care. This study is based on a successful application of Jumpstart Form in the outpatient clinic setting.

ELIGIBILITY:
Inclusion Criteria, Patients: meeting criteria for serious illness (encompassing multiple acute and chronic illnesses) including:

* those used by the Dartmouth Atlas to study end-of-life care in the US: malignant cancer/leukemia, chronic pulmonary disease, coronary artery disease, congestive heart failure, chronic liver disease, chronic renal disease, dementia, diabetes with end-organ damage, and peripheral vascular disease.
* patients over age 65 with markers of frailty: albumin level <3.0 within 48 hours of admission and weight loss of ≥10 pounds in the past year.
* hospitalized patients over age 80.
* English-speaking

Exclusion Criteria, Patients:

* unable to complete informed consent procedures and do not have a legal next of kin
* restricted information status (e.g. prisoners)
* pregnant

Inclusion Criteria, Surrogates:

* involved in the care of an eligible patient as the legal next-of-kin
* English-speaking

Exclusion Criteria, Surrogates:

* unable to complete informed consent procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Engelberg, PhD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Harborview Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee RY, Kross EK, Downey L, Paul SR, Heywood J, Nielsen EL, Okimoto K, Brumback LC, Merel SE, Engelberg RA, Curtis JR. Efficacy of a Communication-Priming Intervention on Documented Goals-of-Care Discussions in Hospitalized Patients With Serious Illness: A Randomized Clinical Trial. JAMA Netw Open. 2022 Apr 1;5(4):e225088. doi: 10.1001/jamanetworkopen.2022.5088. PMID 35363271

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: Usual in-patient hospital care.
Period: Overall Study
Arm/Group | Jumpstart Intervention | Usual Care
Started | 75 | 75
Completed | 75 | 75
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Jumpstart Intervention | Usual Care | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Median (Full Range); unit: years] | 62 [20 to 92] | 60 [23 to 92] | 61 [20 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 39 | 66
  Male | 48 | 36 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 1 | 9
  Not Hispanic or Latino | 67 | 74 | 141
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 9 | 19
  White | 62 | 54 | 116
  More than one race | 2 | 8 | 10
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: Documentation of Goals of Care
Description: Presence of documentation of goals of care discussions in the patient's electronic health record during the index hospitalization
Time Frame: At hospital discharge, an average of 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Jumpstart Intervention | Usual Care
Number analyzed (Participants) | 75 | 75
Participants | 16 | 6
Statistical Analysis 1: Comparison: Jumpstart Intervention vs Usual Care; Test type: Superiority; p = 0.036, Fisher Exact

ADVERSE EVENTS:
Time Frame: Data were collected throughout the index hospital hospitalization, an average of 2 weeks.
Arm/Group | Jumpstart Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 0/75 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-04): https://cdn.clinicaltrials.gov/large-docs/92/NCT03746392/Prot_SAP_000.pdf